CLINICAL TRIAL: NCT02954263
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled, Multiple Ascending Dose Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of TD-1439 in Healthy Subjects
Brief Title: Multiple Ascending Dose Study of TD-1439 in Healthy Adult and Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 0150
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Healthy Adults, Elderly Subjects
Keywords: Multiple ascending dose (MAD)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TD-1439 (Experimental): Capsule formulation
  Interventions: Drug: TD-1439
- Placebo (Placebo Comparator): Capsule formulation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TD-1439
  Arms: TD-1439
Drug: Placebo
  Arms: Placebo

SUMMARY:
Multiple ascending dose study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of TD-1439 in healthy adult and elderly subjects

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) 18 to 32 kg/m2 inclusive
* Women of child bearing potential must have a negative pregnancy test and either abstain from sex or use highly effective methods of birth control
* Women of non-childbearing potential are at least 2 years postmenopausal or are surgically sterile
* Males must abstain from sex or use highly effective methods of birth control
* Negative for HIV, and Hepatitis A, B, and C

Exclusion Criteria:

* Female subjects who are pregnant, lactating, breastfeeding or planning to become pregnant during the study.
* Subjects with a history of angioedema.
* Subject has evidence or history of clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of dosing), hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease.
* Subject has acute illness (gastrointestinal, infection [e.g., influenza] or known inflammatory process)
* Subject has bradycardia
* Subject has hypertension
* Subjects has orthostatic hypotension
* Subjects has orthostatic tachycardia
* Subject has a known personal or family history of congenital long QT syndrome or known family history of sudden death.
* Subject has donated blood or blood components or has had blood loss exceeding 400 mL within the 90 days prior to Screening.
* Additional exclusion criteria apply

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11; Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The number of adverse events by severity, including changes in vital signs, physical examination, laboratory safety tests, and ECGs. | From Day 1 through end of study (Day 25)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of TD-1439 in plasma after multiple doses - peak plasma concentration (Cmax) | Day 1 to 3 days after last dose (Day 17)
PK of TD-1439 in plasma after multiple doses - time to peak plasma concentration (Tmax) | Day 1 to 3 days after last dose (Day 17)
PK of TD-1439 in plasma after multiple doses - time to last measurable concentration (Tlast) | Day 1 to 3 days after last dose (Day 17)
PK of TD-1439 in plasma after multiple doses - area under the plasma concentration vs. time curve from time zero to the last quantifiable concentration (AUC0-t) | Day 1 to 3 days after last dose (Day 17)
PK of TD-1439 in plasma after multiple doses - area under the plasma concentration vs. time curve from time zero to 24 hours postdose (AUC0-24) | Day 1 to 3 days after last dose (Day 17)
PK of TD-1439 in plasma after multiple doses - CL/F (oral plasma clearance) | Day 1 to 3 days after last dose (Day 17)
PK of TD-1439 in plasma after multiple doses - Vz/F (apparent volume of distribution during the terminal phase) | Day 1 to 3 days after last dose (Day 17)
PK of TD-1439 in plasma after multiple doses - t1/2 (half-life) | Day 1 to 3 days after last dose (Day 17)
PK of TD-1439 in urine after multiple doses - Ae (amount excreted in urine) | Day 1 to 3 days after last dose (Day 17)
PK of TD-1439 in urine after multiple doses - Fe (fraction of oral dose excreted in urine) | Day 1 to 3 days after last dose (Day 17)
PK of TD-1439 in urine after multiple doses - Clr (renal clearance) | Day 1 to 3 days after last dose (Day 17)
Pharmacodynamic assessments for plasma atrial natriuretic peptide (ANP) concentrations | The day before dosing (Day -1) to 3 days after last dose (Day 17)
Pharmacodynamic assessments for plasma cyclic guanosine monophosphate (cGMP) concentrations | The day before dosing (Day -1) to 3 days after last dose (Day 17)
Pharmacodynamic assessments for urine cyclic guanosine monophosphate (cGMP) concentrations | The day before dosing (Day -1) to 3 days after last dose (Day 17)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.